CLINICAL TRIAL: NCT02594410
Title: The Efficacy of Renal Artery Stent Combined With Standardized Medical Therapy in Patients With Atherosclerotic Renal Artery Stenosis
Brief Title: Zainidip in Renal Artery Stenosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zhaoke-1503-zanidip
Record Dates: First submitted 2015-10-29; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Stents; Clopidogrel; lercanidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): patients receiving renal artery stenting and anti-hypertension drug for renal artery atherosclerosis
  Interventions: Device: stent; Drug: Aspirine; Drug: Clopidogrel; Drug: Lercanidipine

INTERVENTIONS:
Device: stent — patients receiving renal artery stenting for renal artery atherosclerosis
Drug: Aspirine — 100mg Qd
Drug: Clopidogrel — 75mg Qd
Drug: Lercanidipine — 10-20mg Qd

SUMMARY:
To evaluate the efficacy of renal artery stent combined with standardized medical therapy as treatment for renal artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 - 75
* Diameter of stenosis of renal artery or main branch of renal artery ≥60％. If diameter of stenosis is 60% - 75%, pressure difference between proximal and distal end ≥20 mm Hg (1mmHg=0.133kPa) or Captopril renography positive;
* Systolic blood pressure before taking antihypertensive ≥180mmHg and/or diastolic blood pressure ≥110 mmHg; taking three antihypertensive including one diuretics with systolic blood pressure ≥140mmHg and/or ≥90 mmHg;
* length of ipsilateral kidney is greater than 7.0cm.

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) <30 ml/ (min﹒1.73 m 2) [eGFR (mL/min/1.73 m2) = 186.3 * serum creatinine (mg/dl) -1.154 * Age-0.203 * 0.742 (female)[11];
* unstable condition and unable to tolerate interventional therapy;
* anatomy of renal artery pathology not suitable for interventional therapy;
* allergic to dihydropyridines;
* III degree atrioventricular block
* contrast allergy ;
* any known malignant tumor;
* non-compliant, history of alcoholism or drug abuse.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate | 12 months
Blood pressure | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, China